CLINICAL TRIAL: NCT00783601
Title: A Multicenter, Randomized, Double Blind, Crossover Study Comparing the Effect of MK0524 With Placebo and Concomitant Administration of MK0524 Plus Montelukast in Adult Patients With Chronic Asthma
Brief Title: MK0524 Asthma POC Study (0524-008)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-008; MK0524-008; 2007_614
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Chronic Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Treatment Sequence 1: MK0524 + placebo, MK0524 + montelukast, placebo, placebo, placebo + montelukast
  Interventions: Drug: Comparator: MK0524 + placebo; Drug: Comparator: MK0524 + montelukast; Drug: Comparator: placebo + montelukast; Drug: Comparator: Placebo
- 2 (Experimental): Treatment sequence 2: Placebo, montelukast, placebo, MK0524, MK0524 + montelukast
  Interventions: Drug: Comparator: MK0524 + placebo; Drug: Comparator: MK0524 + montelukast; Drug: Comparator: placebo + montelukast; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: MK0524 + placebo — Two 150 mg MK0524 tablets + one placebo tablet in the matching image of montelukast 10 mg once daily for 3 weeks
Drug: Comparator: MK0524 + montelukast — Two 150 mg MK0524 tablets and one 10 mg montelukast tablet once daily for 2 weeks
Drug: Comparator: placebo + montelukast — Two placebo tablets in the matching image of MK0524 150 mg and one 10 mg tablet montelukast once daily for 2 weeks
Drug: Comparator: Placebo — During the double-blind treatment periods, patients receive either two placebo tablets in the matching image of MK0524 150 mg or one placebo tablet in the matching image of montelukast 10 mg in a crossover manner. During the washout period before the crossover to the opposite treatment sequence, patients receive two placebo tablets in the matching image of MK0524 150 mg and one placebo tablet in the matching image of montelukast 10 mg once daily for two weeks.

SUMMARY:
The purpose of the study is to demonstrate the benefit of MK0524 compared to placebo in patients with chronic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Has symptoms of chronic asthma (shortness of breath, wheezing, chest tightness, etc.) for at least 1 year
* Nonsmoker for at least 1 year with a smoking history of no more than 7 pack-years (i.e., 1 pack per day for 7 years)

Exclusion Criteria:

* Any clinically significant disease of heart, intestinal, kidney, liver, lung or uncontrolled blood pressure
* Any surgery within 4 weeks prior to Visit 1
* Patient is intending to move or vacation for more than 5 days during the study
* Patient is pregnant or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate benefits of MK0524 compared with placebo on Forced Expiratory Volume in 1 second (FEV1) | Last 2 weeks of each treatment period

SECONDARY OUTCOMES:
To determine the benefits of MK0524 as compared with placebo on the key secondary endpoints (Daytime & Nighttime Asthma Symptoms scores | Last 2 weeks of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Philip G, van Adelsberg J, Loeys T, Liu N, Wong P, Lai E, Dass SB, Reiss TF. Clinical studies of the DP1 antagonist laropiprant in asthma and allergic rhinitis. J Allergy Clin Immunol. 2009 Nov;124(5):942-8.e1-9. doi: 10.1016/j.jaci.2009.07.006. Epub 2009 Sep 12. PMID 19748656